CLINICAL TRIAL: NCT00774774
Title: a Randomized Controlled Trial Evaluating the Effectiveness and the Safety of Surgical Masks Wared by the Index Patient for Preventing Secondary Transmission of Influenza A in Households
Brief Title: Face Masks for Preventing Influenza Transmission
Acronym: GRIPMASK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: laurent piazza, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P070160
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2008-09

CONDITIONS: Influenza Human
Keywords: Influenza, human; Masks; Disease Transmission, Horizontal
MeSH Terms: conditions — Influenza, Human | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): No intervention
  Interventions: Device: control
- 1 (Experimental): Mask
  Interventions: Device: Face mask

INTERVENTIONS:
Device: control — Non sterile surgical mask,high filtration "AEROKYN",type 2 with eardrop
  Arms: 2
Device: Face mask — Non sterile surgical mask, high filtration "AEROKYN", type 2 with eardrop Masks will be worn at home by the patient over a period of 5 days following inclusion, whenever a member of the household will attend the same room or in other confined space (eg car), and changed after 3 hours of consecutive use or sooner if they are tor
  Masks will not be worn:
  * during the night,
  * when the patient is alone in the room. Moreover, for all households, an incentive in nocturnal isolation of index-patient will be recommended
  Arms: 1

SUMMARY:
This work aims to measure the effectiveness of face mask worn by a patient with flu to avoid transmission to other persons in the household.

DETAILED DESCRIPTION:
Background. Non pharmaceutical interventions, and in particular the wearing of face masks, could play a role in controlling the transmission of influenza in the early stages of the epidemic. In the French pandemic plan, surgical masks are recommended in contagious patients in wards. The effectiveness of such masks in preventing transmission of influenza A virus is unknown. Our project aims to assess the preventive efficacy and tolerance of surgical mask.

The primary objective is to measure the decrease of the number of secondary cases of flu in households where the index case will wear a surgical mask during its period of infectiousness (5 days), compared to households where the index case will not be subject to this intervention. Secondary objectives are: (1) to study the feasibility and tolerance of wearing a mask continuously during the period of viral shedding; (2) virological description of infection spreading among household contacts based on virological collections.

ELIGIBILITY:
Inclusion Criteria:

Patient seeking medical advice for:

* For symptoms less than 48 hours, combining fever> = 37.8 ° C and a cough,
* during the period of a seasonal influenza epidemic (as defined by the Sentinel network)
* Older than 5 years
* And living in a household size between 3 to 8..
* The patient is the first case in the household (index patient). The patient has a positive rapid influenza A test.
* Informed consent.
* Affiliation to the social security.

Exclusion Criteria:

* When concomitant influenza cases are known in other householders
* When the patient is suffering from asthma or COPD (ongoing treatment):
* Hospitalization.
* Treatment by a neuraminidase inhibitor.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The number of household contacts who will develop within 7 days of the inclusion of the index patient a respiratory syndrome defined by fever> = 37.8 ° C and a cough or a sore throat. | during the study

SECONDARY OUTCOMES:
clinical events in all household members on the entire monitoring period (21 days). | 21 days
Adverse events related to wearing a mask - a safety issue. | during the study
Number of days of wearing a mask, number of masks used. | during the study
Drug-consumption, in particular antibiotics | during the study
Sick-leave from work (for adults contacts), or from school (for children of school age). | during the study
Quality of life in the index patient. | during the study
Infection with influenza virus at different time, among all household members. | during the study
Quantification of viral load in patients infected. | during the study
Characterization of viruses isolated (sub-type and sequence of the portion of HA1 gene for haemagglutinin). | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice CARRAT, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Saint Antoine, Paris, France

REFERENCES:
- [Result] Sies H, Akerboom TP, Tager JM. Mitochondrial and cytosolic NADPH systems and isocitrate dehydrogenase indicator metabolites during ureogensis from ammonia in isolated rat hepatocytes. Eur J Biochem. 1977 Jan;72(2):301-7. doi: 10.1111/j.1432-1033.1977.tb11253.x. PMID 13998
- [Derived] Canini L, Andreoletti L, Ferrari P, D'Angelo R, Blanchon T, Lemaitre M, Filleul L, Ferry JP, Desmaizieres M, Smadja S, Valleron AJ, Carrat F. Surgical mask to prevent influenza transmission in households: a cluster randomized trial. PLoS One. 2010 Nov 17;5(11):e13998. doi: 10.1371/journal.pone.0013998. PMID 21103330